CLINICAL TRIAL: NCT06453369
Title: A Novel Vertical Y-shaped Tunnel Approach Versus Modified Coronally Advanced Tunnel Technique, for The Treatment of Miller Class I Gingival Recession - Randomized Clinical Trial
Brief Title: A Novel Vertical Y-shaped Tunnel Approach Versus Modified Coronally Advanced Tunnel Technique, for The Treatment of Miller Class I Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Aslam Ashraf Mogahed, principle investigator. Aslam Ashraf Mogahed, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-2022
Record Dates: First submitted 2024-05-07; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Gingival Recession
Keywords: gingival recession; Modified tunnel technique; tunnel technique; connective tissue graft; minimally invasive; root coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- root coverage using novel Y shaped Tunnel with Connective tissue graft (Experimental): Sulcular incision will be performed using 15c blade . Micro-periosteal elevator will be used to elevate vertical full thickness tunnel starting coronally from the gingival sulcus and directed apically. Micro periosteal elevator will be used to elevate the buccal aspect of both mesial and distal papillae of the affected tooth. CTG will be prepared and inserted into the coronal tunnel aperture using blunt instrument to facilitate intrusion of graft into tunnel. CTG will be inserted into the tunnel up to the apical level leaving a coronal part to completely cover the recession defect. Finally single interrupted suture will be used to secure the coronal exposed part of the CTG followed by sling suture fixation of the gingival flap with that of CTG. The donor CTG will be stabilized to the underlying connective tissue interproximally using 5.0 sutures.
  Interventions: Procedure: Y shaped Tunnel with Connective tissue graft
- root coverage using MCAT with Connective tissue graft (Active Comparator): The tunnel will be prepared with a full-thickness incision up to MGJ and as a split-thickness beyond MGJ using tunneling instruments to obtain a tension-free tunnel, allowing the insertion of the CTG, a delicate incision is performed at the level of interdental papillae and raised without detaching the tip of the papillae. The papillary regions will be detached in their buccal aspects. The adjacent papillae of the neighboring teeth will be involved in the preparation to ensure a coronal positioning of the flap. After planing, the graft will be inserted into the tunnel by a specific suture technique. The first suture will be inserted through the most distal recession part and the needle exits in the most medial part of the recession, second suture will be placed at the opposite side and the needle exits at the same medial recession. The buccal flap will be advanced coronally to cover CTG and secured with sling sutures. The donor CTG will stabilized to the underlying CT interproximally.
  Interventions: Procedure: Y shaped Tunnel with Connective tissue graft

INTERVENTIONS:
Procedure: Y shaped Tunnel with Connective tissue graft — Sulcular incision followed by Micro-periosteal elevator will be used to elevate vertical full thickness tunnel starting coronally from the gingival sulcus and directed apically. CTG will be prepared and inserted into the coronal tunnel aperture using blunt instrument to facilitate intrusion of graft into tunnel. CTG insurted into the tunnel up to the apical level leaving a coronal part to completely cover the recession defect. Finally single interrupted suture will be used to secure the coronal exposed part of the CTG followed by sling suture fixation of the gingival flap with that of CTG. The donor CTG will be stabilized to the underlying connective tissue interproximally using 5.0 sutures.

SUMMARY:
Recent plastic procedures have provided satisfactory results in the treatment of gingival recession but there is, presently, a greater need for procedure that cause less surgical morbidity as also provide improved results. In this study we propose a novel vertical tunnel technique as a minimally invasive approach (Vertical Y-shaped Tunnel Approach) and evaluate clinical results in comparison to CAMT, both using CTG. The novel technique allows stability of the graft, maximum coronal vascularity and minimum soft tissue reflection.

DETAILED DESCRIPTION:
The tunnel technique is an approach that optimizes esthetics and predictability because of its ability to avoid releasing critical papillae and maintaining a high level of vascularity at the surgical site to support the grafts. The tunnel technique has a minimally invasive nature since the interdental papillae are left intact and vertical incisions are not performed which results in better esthetics. This technique entailed the placement of a connective tissue graft in the tunnel. Complete graft coverage is not mandatory as long as the graft dimensions are sufficient to ensure its survival. Avoiding detachment of the highly fragile interdental soft tissue can minimize the risk of losing papilla height in critical esthetic areas, avoid scar formation, maximize the papillary and lateral blood supply to the underlying graft and better stabilize the graft for optimal wound healing Recent plastic procedures have provided satisfactory results in the treatment of gingival recession but there is, presently, a greater need for procedure that cause less surgical morbidity as also provide improved results. In this study we propose a novel vertical tunnel technique as a minimally invasive approach (Vertical Y-shaped Tunnel Approach) and evaluate clinical results in comparison to CAMT, both using CTG. The novel technique allows stability of the graft, maximum coronal vascularity and minimum soft tissue reflection.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years old.
2. The presence of Miller's class I gingival recession (25).
3. Recession defect on maxillary incisors, maxillary and mandibular canines, or premolars.
4. Absence of a history of periodontal surgery at the involved sites in the last 12 months.
5. History of compliance with oral hygiene instructions and periodontal recall.
6. Sufficient palatal donor tissue thickness (> 2mm).
7. Clearly identifiable cemento-enamel-junction (CEJ)

Exclusion Criteria:

1. Patients with systemic illness known to affect the outcome of periodontal therapy, including diabetes, immune deficiencies, etc (26).
2. Pregnant and lactating women
3. Current use of any form of tobacco.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-02-04 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
percentage of root coverage | 1 month, 3 and 6 months
  Percentage root coverage (%RC): calculated as ([RD preoperative - RD postoperative]/RD preoperative) × 100%.

SECONDARY OUTCOMES:
Complete root coverage (CRC) | 1 month, 3 and 6 months
  The number of sites that resulted in 100% root coverage.
Recession Depth (RD) | 1 month, 3 and 6 months
  Measured in millimeters from the gingival margin at the midbuccal aspect of the root, to the CEJ or relative CEJ.
Recession width (RW) | 1 month, 3 and 6 months
  The horizontal distance between the bilateral gingival margins at the height of the CEJ. (mm)
Probing depth (PD) | 6 months
  Measured in millimeters from the gingival margin to the base of the periodontal sulcus at 6 sites per tooth. (baseline and after 6 months)
Clinical attachment level (CAL) | 6 months
  Measured in millimeters from CEJ or relative CEJ to the base of the periodontal sulcus at 6 sites per tooth. (after 6 months)
Width of the keratinized tissue (KTW) | 1 month, 3 and 6 months
  Measured in millimeters at midbuccal aspect of the tooth from the gingival margin to the mucogingival junction.
Gingival Thickness (GT) | 6 months
  Measured in millimeters at the mid-buccal of the gingiva and 2 mm apical the gingival margin at the attached gingiva or the alveolar mucosa using a #15 endodontic reamer with a silicon disk stop.
Plaque index (PI) | 1 month, 3 and 6 months
  Is used for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin.
Gingival index (GI) | 1 month, 3 and 6 months
  GI is measured according to Loe and Sillness and scored on a scale of 0 to 3.
Pain index (PN) | 1 month, 3 and 6 months
  Pain is recorded on a horizontal pain scale of 0-10, Pain index to be recorded by the patients at 9 am, 3pm, and 9 pm from the day of the surgery and for 3 weeks post-treatment.
Professional esthetic evaluation and patient-reported satisfaction | 6 months
  The esthetic outcome will be assessed post-operatively after 6 months by an independent second examiner (MS), who is blinded to the treatment assignment, in accordance with RES (30). The evaluation will be based on comparing digital photographs.
  Five variables were assessed:
  1. the level of gingival margin (GM);
  2. marginal tissue contour (MTC);
  3. soft tissue texture (STT);
  4. muco-gingival junction alignment (MGJ); and
  5. gingival color (GC). A score of 0, 3, or 6 will be used for evaluation of GM, whereas a score of 0-1 will be used for each of the other variables. The ideal esthetic score will be 10.

CONTACTS AND LOCATIONS:
Overall Officials: Aslam Ashraf Mogahed, BDs, Principal Investigator — O6U
Locations (1):
- 6 October university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided